CLINICAL TRIAL: NCT06523517
Title: A Single-center, Single-arm, Prospective Clinical Study to Evaluate the Efficacy and Safety of Eliglustat in Chinese Pediatric Patients (≥12 to <18 Years Old) With Gaucher Disease Type 1 and Type 3
Brief Title: Efficacy and Safety of Eliglustat in Chinese Pediatric Patients With Gaucher Disease Type 1 and Type 3
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Peking Union Medical College Hospital (Other)
Responsible Party: Principal Investigator, Bing Han, Professor, Peking Union Medical College Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Eliglustat
Record Dates: First submitted 2024-07-18; First posted 2024-07-26 (Actual); Last update posted 2024-07-26 (Actual); Status verified 2024-07

CONDITIONS: Gaucher Disease
Keywords: Eliglustat
MeSH Terms: conditions — Gaucher Disease | interventions — eliglustat

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- treatment group (Experimental): Eliglustat Tartrate Capsules, either 42 mg or 84 mg taken orally twice a day for 52 weeks.
  Interventions: Drug: Eliglustat Tartrate Capsules

INTERVENTIONS:
Drug: Eliglustat Tartrate Capsules — The initial dose is 42 mg taken orally twice a day. After 2 weeks of treatment, if the blood trough concentration is less than 5 ng/mL, the dose will be increased to 84 mg taken orally twice daily.

SUMMARY:
Primary Objective:

Evaluate the efficacy and safety of eliglustat in Chinese pediatric patients (≥12 to <18 years old) with Gaucher disease type 1 and type 3.

Secondary Objective:

Evaluate the quality of life in Chinese pediatric patients (≥12 to <18 years old) with Gaucher disease type 1 and type 3 treated with eliglustat.

ELIGIBILITY:
Inclusion Criteria:

* The patient is ≥12 to <18 years old at the time of informed consent.
* The patient is diagnosed with Gaucher disease based on the following criteria:

  1. Glucocerebrosidase (GBA) activity reduced to ≤30% of the lower limit of normal, or
  2. GBA activity reduced by >30% of the lower limit of normal, but confirmed by glucocerebrosidase (GBA) genotype.
* Postmenarchal female patients must have a documented negative pregnancy test prior to enrollment and throughout the study.
* Patients must have been receiving enzyme replacement therapy (ERT) for a minimum of 24 months at a monthly dose equivalent to 30 U/kg to 130 U/kg of enzyme, with treatment ongoing at the time of enrollment. Patients must meet pre-specified treatment goals defined as:

  1. Hemoglobin levels: ≥11.0 g/dL for females and ≥12.0 g/dL for males;
  2. Platelet count ≥100,000/mm³;
  3. Spleen volume <10.0 multiples of normal (MN);
  4. Liver volume <1.5 MN.
* After explaining and discussing all relevant aspects of the study with the patients and their guardians, patients and their guardians must voluntarily sign the written informed consent form approved by the institutional ethics committee.
* Cytochrome P450 2D6 (CYP2D6) genotype testing shows extensive metabolizers (EMs) or intermediate metabolizers (IMs).
* Patients agree to avoid consuming grapefruit and grapefruit juice.
* Patients agree to discontinue medications listed as contraindicated for concomitant use.
* Participants must be able to cooperate fully as determined by the Principal Investigator to be eligible for the study.

Exclusion Criteria:

* Underwent substrate reduction therapy (SRT) for GD or received miglustat treatment within 12 months prior to enrollment.
* Underwent partial or total splenectomy prior to enrollment or experienced active, clinically significant splenic infarction within the previous 12 months.
* The patient is transfusion-dependent; has a history of esophageal varices or liver infarction; elevated liver enzymes; significant congenital cardiac defect; coronary artery disease; left-sided heart failure; clinically significant arrhythmias; or conduction defects such as Type 2 second-degree or third-degree atrioventricular (AV) block, complete bundle branch block, prolonged QTc interval, or sustained ventricular tachycardia (VT).
* Presence of significant comorbidities, as determined by the Principal Investigator, which may affect study data or confound study results (e.g., malignancies, primary biliary cirrhosis, autoimmune liver disease, pulmonary complications, cardiac structural or functional abnormalities, etc.).
* The patient with any clinically significant disease other than GD.
* Experienced severe bone disease such as new-onset bone crises or fractures within 12 months prior to enrollment.
* The patient has received an investigational product within 30 days prior to enrollment.
* The patient has a known hereditary galactose intolerance, Lapp lactase deficiency, glucose galactose malabsorption, or is a CYP2D6 ultra-rapid metabolizer or indeterminate metabolizer.
* The patient is currently receiving erythropoiesis-stimulating agents (e.g., erythropoietin) or long-term systemic corticosteroid therapy, or received such treatment within 6 months prior to enrollment.
* Positive hepatitis B surface antigen (HBsAg) test results with detectable hepatitis B virus DNA load; positive hepatitis C virus (HCV) antibody with confirmation by HCV RNA polymerase chain reaction (PCR) testing; and positive human immunodeficiency virus (HIV) antibody at screening.
* Presence of non-GD-related hemolytic anemia (such as due to iron, folate, and/or vitamin B12 deficiency or infection/immune-mediated causes) at screening. Patients with folate deficiency, vitamin B12 deficiency-related anemia, or iron deficiency-related anemia at screening are ineligible for study enrollment and will be considered screening failures. Patients may receive treatment for underlying conditions and be re-screened at the discretion of the Principal Investigator.
* The patient and their guardian are unable to comprehend the nature, scope, and potential consequences of the study.
* The Principal Investigator determines that the patient is unsuitable for participation in the clinical trial based on the subject's overall condition.

Ages: 12 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 5 (Estimated)
Dates: Start 2024-08-01 (Estimated); Primary Completion 2025-07-31 (Estimated); Study Completion 2025-07-31 (Estimated)

PRIMARY OUTCOMES:
Changes in hemoglobin level | Baseline, Weeks 13, 26, 39 and 52
  Absolute change from baseline for hemoglobin (g/dL)
Changes in platelet count | Baseline, Weeks 13, 26, 39 and 52
  Percent change from baseline for platelet count
Changes in spleen volume | Baseline, Weeks 26 and 52
  Percent change from baseline for spleen volume
Changes in liver volume | Baseline, Weeks 26 and 52
  Percent change from baseline for liver volume
Changes in Lyso-GL1 level | Baseline, Weeks 13, 26, 39 and 52
  Percent change from baseline for Lyso-GL1 level
Skeletal improvement | Baseline, Weeks 26 and 52
  Proportion of patients with improvement in skeletal disease
Assessment of pharmacokinetic (PK) parameter of eliglustat: Cmax | Baseline, Weeks 2, 13, 26 and 52
  Peak concentration (Cmax) of eliglustat in plasma (ng/mL)
Assessment of pharmacokinetic (PK) parameter of eliglustat: Ctrough | Baseline, Weeks 2, 13, 26 and 52
  Trough concentration (Ctrough) of eliglustat in plasma (ng/mL)
Adverse events | Up to Week 52
  Number of adverse events in pediatric patients

SECONDARY OUTCOMES:
Changes in Quality of Life | Baseline and Week 52
  Health-related quality of life will be measured by the Pediatric Quality of Life Inventory™ (PedsQL™) questionnaires

CONTACTS AND LOCATIONS:
Overall Officials: Bing Han, Principal Investigator — Peking Union Medical College
Locations (1):
- Peking union medical college hospital, Beijing, China

IPD SHARING:
Plan to Share IPD: No